CLINICAL TRIAL: NCT06724874
Title: The Effect of Online Web-Based Deep Relaxation Exercise Applied to Pregnant Women on Maternal Fetal Attachment and Pregnancy Perception: A Randomized Controlled Trial
Brief Title: Online Web-Based Deep Relaxation Exercise Applied to Pregnant Women on Maternal Fetal Attachment and Pregnancy Perception
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Çankırı Karatekin University (Other)
Responsible Party: Principal Investigator, Nilay Gökbulut, Assist. Prof. Dr., Çankırı Karatekin University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KARATEKIN UNIVERSITY
Record Dates: First submitted 2024-12-05; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Maternal Fetal Attachment Pregnancy Perception; Pregnancy Perception

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention)
- Web-based deep relaxation exercise (Experimental)
  Interventions: Other: Web-Based Deep Relaxation Exercise

INTERVENTIONS:
Other: Web-Based Deep Relaxation Exercise — Web-based deep relaxation exercise videos have been prepared online. Each video lasts approximately 20-25 minutes. The 4-week applications will be sent to pregnant women one video each week and they will be asked to continue the exercises at home 4 times a week.
  Arms: Web-based deep relaxation exercise

SUMMARY:
This study was planned as a pre-test post-test randomized controlled study in order to determine the effects of an online web-based deep relaxation exercise applied to pregnant women on maternal-fetal attachment and pregnancy perception. The study is planned to be conducted with pregnant women reached through social media (such as Facebook, Messenger, Instagram). The study is planned to be conducted between December 15, 2024 and June 15, 2025. The universe of the study will consist of pregnant women who volunteer to participate in online deep relaxation exercises and share their contact information. When the power analysis was performed, the sample size was calculated as a total of 80 pregnant women (40 experimental, 40 control), assuming that the web-based deep relaxation exercise applied would increase the mean maternal-fetal attachment score (72.25±7.16) (Güney and Uçar, 2019) by four and a half points at a 5% error level, a two-sided significance level, a 95% confidence interval, and an 80% ability to represent the universe (https://www.stat.ubc.ca/~rollin/stats/ssize/n2.html). Pregnant women to be included in the groups will be selected from the relevant population using the improbable random sampling method.

ELIGIBILITY:
Inclusion Criteria:

* Women with internet access,
* Women expecting a single baby,
* Women whose pregnancy is 12-24 weeks

Exclusion Criteria:

* Women with a history of physical and/or psychological illness and those taking any psychiatric medication
* Women who answered the survey questions incompletely.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-12-15 (Estimated); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Effect of online web-based deep relaxation exercise applied to pregnant women on maternal-fetal attachment | Four months

SECONDARY OUTCOMES:
The effect of online web-based deep relaxation exercise applied to pregnant women on pregnancy perception | Four months

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared, because before starting the research, pregnant women who will participate in the research, as they will be guaranteed that their personal information will be kept completely confidential and will only be used for this research purpose.

REFERENCES:
- [Background] Kumcağız H, Ersanlı E, Murat N. The Development of a Self-perception of Pregnants Scale and its Psychometric Features.Journal of Psychiatric Nursing 2017;8(1):23-31
- [Background] Golbasi Z, Ucar T, Tugut N. Validity and reliability of the Turkish version of the Maternal Antenatal Attachment Scale. Jpn J Nurs Sci. 2015 Apr;12(2):154-61. doi: 10.1111/jjns.12052. Epub 2014 Jun 24. PMID 24962076
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/24962076/
- Available data/document: Individual Participant Data Set — https://www.stat.ubc.ca/~rollin/stats/ssize/n2.html